CLINICAL TRIAL: NCT06126445
Title: Dental Plaque Removal Efficacy Evaluation and Comparison of Electric Toothbrush and Manual Toothbrush
Brief Title: Single Brushing Plaque Removal Efficacy of a Battery-powered Toothbrush and a Manual Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ST-23-U34
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Plaque, Dental
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: single use, examiner blinded, randomized, two-period, cross-over
Who Masked: Investigator
Masking Description: Examiner blinded to toothbrush used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Battery operated toothbrush (Active Comparator): battery operated toothbrush
  Interventions: Device: Battery operated toothbrush
- Manual toothbrush (Active Comparator): Manual toothbrush
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Battery operated toothbrush — Device on plaque removal efficacy
  Arms: Battery operated toothbrush
Device: Manual toothbrush — Device on plaque removal efficacy
  Arms: Manual toothbrush

SUMMARY:
To evaluate and compare the plaque removal efficacy of a battery-powered toothbrush and a manual toothbrush following a single brushing.

DETAILED DESCRIPTION:
This is a single use, examiner blinded, randomized, two-period, cross-over, IRB-approved research study evaluating the single-use plaque removal efficacy of a new battery-operated toothbrush and a marketed manual toothbrush. This study will accept up to 64 subjects, 18-65 years of age, in anticipation that 60 subjects will complete the study. Qualified subjects with sufficient plaque, according to Rustogi Modified Navy Plaque Index (RMNPI) will be randomly assigned to one of two sequence treatment groups.

After the pre-brushing plaque evaluation at each of the evaluation visits, subjects will brush with the assigned toothbrush and toothpaste provided for timed brushing under supervision, in front of mirror.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided a signed and dated informed consent document indicating that you have been informed of all pertinent aspects of the study before any assessments are performed. You will receive a copy of the signed informed consent.
2. Be between 18 and 65 years of age (inclusive), male or female.
3. Able to brush their own teeth on a daily basis.
4. Be in good health based on medical history review by the Principal Investigator.
5. Have a minimum of at least 18 natural, gradable teeth.
6. Have a mean full-mouth pre-brushing plaque score (Rustogi Modification of the Navy Plaque Index, RMNPI) of ≥ 0.50 at evaluation visits 2 & 3.
7. Have agreed to refrain from use of all oral hygiene products (i.e. floss, mouthwash, etc.), other than the toothbrush and toothpaste supplied, for the duration of the study including the acclimation periods.
8. Have agreed to refrain from all oral hygiene and chewing gum for approximately 12-16 hours and refrain from eating, drinking, smoking and chewing gum for approximately 4 hours prior to Visits 2 & 3.
9. Have agreed not to have a dental prophylaxis or any other elective, non-emergency dental procedures (other than those provided during the study) any time during the study.
10. Approximately 50% of subjects will be regular electric toothbrush users and 50% of subjects will be regular manual toothbrush users.
11. Have agreed to comply with the conditions and schedule of the study.

Exclusion Criteria:

1. Have any physical limitations or restrictions which might preclude normal tooth brushing.
2. Have to be premedicated prior to dental treatment.
3. Have evidence of poor oral hygiene or rampant dental caries or calculus deposits that may interfere with plaque assessments.
4. Have evidence of major oral hard or soft tissue lesions or trauma at Baseline.
5. Have fixed or removable orthodontic appliances.
6. Have received a dental prophylaxis within a month prior to Visit 1.
7. Have a history of a significant adverse event, allergy, or irritation that was due to oral hygiene products.
8. Have participated in another dental research study within 4 weeks prior to Visit 1.
9. Therapy with any medications, currently or within the last 28 days, which might interfere with the outcome of the study by affecting tissue condition, or salivation, particularly chronic therapy or long-term use, as determined by the investigator.
10. Existing serious medical condition or transmittable disease as determined by the Principal Investigator after review of the medical history form. These will include but not be limited to, hepatitis, tuberculosis, AIDS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Within-Treatment Whole-Mouth Differences (vs Baseline) - Plaque removal | up to 2 weeks
  Mean Change from baseline (pre-brushing to post-brushing) in plaque score after single supervised use based on all surfaces of the whole mouth measured. Scale used is Rustogi Modification of the Navy Plaque Index (RMNPI). Up to 504 sites scored in the mouth, with each score a 0 or 1, and subject scores an average over all sites measured. Minimum score of 0 and maximum score of 1. For each timepoint, a larger score means more plaque. For reduction from baseline, a larger score means a greater reduction in plaque.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Qaqish, Study Director — All Sum Research Center Ltd.
Locations (1):
- All Sum Research Center Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No